## The Effect of Surgeon Emotional Support on Treatment Choice for Low-Risk Thyroid Cancer

version 10/22/2021

NCT05132478

You are eligible to participate in the study! Please read the information below before proceeding to the study. If you have any questions, please contact the study team.

The CHOiCES Study team led by Corrine Voils, PhD at the University of Wisconsin-Madison and Susan Pitt, MD, MPHS at the University of Michigan invites you to participate in a research study. The purpose of this study is to understand how communication from a surgeon affects patients' treatment choices. We want to improve the way patients and doctors make choices together to ensure patients' goals are met. We expect to enroll about 120 people with benign thyroid nodules in this study.

## If you participate, you will:

- Answer survey questions about yourself, your medical history, your thoughts on thyroid cancer, and your emotional state
- Be assigned by chance (a process called "randomization") to watch one of two videos depicting a surgeon-patient discussion about treatment options for thyroid cancer
- Answer questions about the video, including what treatment you would choose if you were the patient in the video, and your feelings and reactions to the video

Study participation should take 15 to 20 minutes. Completing the study in one sitting is very important. Please complete the study in a quiet place where you can concentrate, and use a tablet or computer rather than your phone. You will earn \$40 after completing the entire study.

Participation in this study is voluntary. You can skip any survey questions that you do not want to answer. Even if you start the study, you are not required to complete it. Psychological risks are minimal, including the potential for experiencing stress or discomfort, and relate to imagining what you would do if you had a diagnosis of thyroid cancer.

Some questions you will complete in this study ask about symptoms of emotional distress such as anxiety. We are using the questions for research purposes only, not to diagnose mental health issues. We will not disclose the results to you. If you are experiencing emotional distress, you should contact your physician or other health care provider, such as a mental health professional, or visit mentalhealth.gov for a list of resources.

Protected health information (PHI) is information about your physical or mental health that includes your name or other information that can identify you. For this study, we will only use your answers to the survey, which include questions related to your health. When you complete this study, you give researchers permission to use your answers now and in the future. However, you can choose to take back your authorization for researchers to use your health information. To take back your authorization, you may contact us at any time.

All of your answers are confidential and will be shared only with the research team, including researchers at the University of Michigan. Contact information will be kept confidential and will only be used for mailing payment for participation.

We will keep your data for an indefinite period of time, meaning we have no plans of ever destroying them. Keeping data for future research is called "banking." The banked data will be kept in a secure location for use by researchers. Your data may be shared for future research but only after identifiable private information such as your name are removed. The data may be shared with other researchers at the University of Wisconsin-Madison and outside the University. Outside researchers may be at other universities, private companies, or other kinds of organizations. Banked data will not be shared with your health care providers.

A description of this study will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

If you have any questions about your rights as a research participant or have complaints about the research study or study team, contact the Anonymous Human Research Protection Hotline, which works with research participants to address concerns about research participation and assist in resolving problems. They can be reached at (608)890-1273, (833)652-2506 (toll free), or hrpp@research.wisc.edu.

If you have questions about the study after reading this page, please contact the study coordinator Kyle Bushaw at choicestudy@surgery.wisc.edu or (608)265-2904 before proceeding to the next page. If you do not want to participate or be contacted about the study again, please contact us to let us know.

By clicking to the next page, you indicate your consent to participate in this study.